CLINICAL TRIAL: NCT01841996
Title: A Phase 1 Randomized, Double-Blind, Vehicle-Controlled, Multiple-Dose Study of the Safety, Absorption and Systemic Pharmacokinetics of ME1111 Topical Agent Applied to All Toenails of Adult Moderate to Severe Onychomycosis Patients for 28 Days
Brief Title: Pharmacokinetics and Safety Study of ME1111 in Moderate to Severe Onychomycosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ME1111-1
Record Dates: First submitted 2013-04-18; First posted 2013-04-29 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ME1111 solution (Experimental)
  Interventions: Drug: ME1111 solution
- Vehicle Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Solution

INTERVENTIONS:
Drug: ME1111 solution — Once a day for 28 days
  Arms: ME1111 solution
Drug: Vehicle Solution — Once a day for 28 days
  Arms: Vehicle Solution

SUMMARY:
This study is Randomized, Double-Blind, Vehicle-Controlled, Multiple-Dose Study.

The purpose is to determine the safety, tolerability, systemic exposure and pharmacokinetics of ME1111 after repeated daily topical application of ME1111 in a maximal use setting in adults with distal subungual onychomycosis of the toenails.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race and between the ages of 18 and 70 inclusive
2. Clinically diagnosed onychomycosis of the target nail
3. Presence of moderate to severe distal subungual onychomycosis
4. A positive potassium hydroxide(KOH) microscopy test result
5. A positive fungal culture for a dermatophyte
6. Females of childbearing potential must be using a highly effective method of birth control and be willing to remain on the same method of birth control throughout the study
7. Good general health as determined by the Investigator based on the subject's medical history and physical examination

Exclusion Criteria:

1. Clinical significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize subject's safety
2. Subjects with a history of diabetes mellitus
3. Unwilling to refrain from the use of nail cosmetics such as clear and/or colored nail solutions
4. Females who are nursing, pregnant, or planning a pregnancy during the study
5. Failure to complete the specified washout period(s) for the following topical medications: Antifungals drugs within 4 weeks; Anti-inflammatory drugs, corticosteroids, immunomodulators within 2 weeks
6. Failure to complete the specified washout period(s) for the following systemic medications: Corticosteroids within 2 weeks; Antifungals for treatment of onychomycosis or any antifungal with known activity against dermatophyte within the previous 24 weeks or 5 half-lives of the drug, whichever is longer; Immunomodulators within 4 weeks
7. History of cardiac disease and cardiac arrhythmic activity, or prolonged QT interval
8. Received treatment for any type of cancer within the last 6 months
9. History of any significant disease or disorder that might put subjects at risk by participating in study or influence results of study
10. Nail or anatomic abnormalities of the toe
11. Positive test for HIV, Hepatitis B or Hepatitis C
12. History of street drug or alcohol abuse
13. Donated or lost blood or participated in a clinical study which involved the withdrawal of a large volume of blood (500 mL or more), within the last 6-week
14. Participated in any other trial of an investigational drug or device within 30 days or 5 half-lives of the investigational drug or participation in a research study concurrent with this study
15. Unable to communicate or cooperate with the Investigator due to comprehension, mental development, or impaired cerebral function
16. Presence of any underlying disease that the Investigator deems uncontrolled, and poses a concern for the subjects safety while participating on the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The number of adverse events observed throughout the study period. | from Baseline to Day 57
Application site reactions will be evaluated using categorical scales for signs and symptoms throughout the study period. | from Baseline to Day 57
Area under the plasma concentration of ME1111 will be assessed based on the analysis of blood samples over 24 hours | Day 1, 28
Urinary excretion rate will be assessed based on the analysis of urinary samples over 24 hours | Day 1, 28
Plasma trough levels of ME1111 | Day 4, 8, 15, 22, 25, 43, 57

SECONDARY OUTCOMES:
Area under the nail concentration of ME1111 | Day 2, 15, 29, 57
The proportion of subjects who achieve negative KOH microscopy testing results | Day 29, 57
The proportion of subjects who achieve negative fungal culture results | Day 29, 57
The change from baseline in linear toenail growth at Days 29 and 57 will be analyzed | Day 1, 29, 57

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuharu Egawa, Study Chair — Meiji Seika Pharma Co., Ltd.
Locations (2):
- United States (2):
  - Austin, Texas
  - College Station, Texas